CLINICAL TRIAL: NCT01858051
Title: Bolus vs. Divided Cholecalciferol Dosing to Optimize Perioperative Vitamin D Status for Joint Replacement Surgery
Brief Title: Vitamin D Status in Lower Extremity Joint Replacement Surgery Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bio-Tech Pharmacal, Inc. (Industry)
Responsible Party: Principal Investigator, Sadeq A. Quraishi, Assistant Professor of Anaesthesia, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013P001071
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Hypovitaminosis D
Keywords: Vitamin D; Perioperative immune regulation; LL-37; Hospital-acquired infection; Surgical site infections
MeSH Terms: conditions — Vitamin D Deficiency; Cross Infection; Surgical Wound Infection | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cholecalciferol Bolus Dose (Active Comparator): 70 patients will receive a bolus pre-operative oral dose of 150,000 IU cholecalciferol 3-7 days before surgery
  Interventions: Dietary Supplement: Cholecalciferol
- Cholecalciferol Divided Dose (Active Comparator): 70 patients will receive an oral 100,000 IU cholecalciferol dose 3-7 days before surgery and an additional oral 50,000 IU cholecalciferol dose on post-operative day 1
  Interventions: Dietary Supplement: Cholecalciferol
- Sugar Pill (Placebo Comparator): 35 patients will receive a placebo pill orally 3-7 days before surgery
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cholecalciferol
  Arms: Cholecalciferol Bolus Dose; Cholecalciferol Divided Dose
Dietary Supplement: Placebo
  Arms: Sugar Pill

SUMMARY:
In the United States, ~1 million elective hip or knee replacement surgeries are performed annually. With estimated surgical site infection (SSI) rates as high as 2.5%, this represents ~25,000 patients at risk of potentially avoidable morbidity following lower extremity joint replacement surgery. Although SSIs only account for 20% of all HAIs, they are a major risk factor for prosthetic joint infections (PJIs). Furthermore, UTIs have also been identified as an independent risk factor for infections of implanted hardware.

In general, the majority of PJIs become apparent within 3 months of hardware implantation, but deep infections may not be evident for up to one year after surgery. Hardware infections result in delayed healing, repeated surgical interventions, and long-term antibiotic therapy. PJIs are associated with an average increase in hospital LOS by 14 days, additional expenditures of up to $50,000 per infected joint, and a doubling of the mortality rate compared to uninfected lower extremity joint replacements.

Recent work from our group suggests that vitamin D insufficiency may be a risk factor for perioperative HAIs. The prevalence of vitamin D insufficiency is approximately 40% in elective joint replacement surgery patients, and perioperative 25(OH)D levels drop 30-40% in the setting of surgical stress, remaining 20% below baseline up to 3 months after surgery. To date, perioperative vitamin D optimization strategies have not been reported. Therefore, our goal is to study the effect of a single (pre-operative) versus a divided (pre-operative and on post-operative day 1) dose of cholecalciferol on perioperative vitamin D status in patients scheduled for elective hip or knee joint replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥18 years
* English or Spanish speaking
* Scheduled for preoperative clinic assessment
* Scheduled to have elective hip or knee joint replacement surgery
* Not taking more than 1000 IU of either cholecalciferol or ergocalciferol daily

Exclusion Criteria:

* Unable to provide consent
* Inability to comply with study protocol
* History of anemia (hematocrit <25%)
* History of renal stones or hypercalcemia
* Conditions that can cause hypercalcemia (e.g. metastatic cancer, sarcoidosis, myeloma)
* Medications that affect vitamin D metabolism (e.g. anti-epileptics, tuberculosis medication)
* Already enrolled or planning to enroll in a research study that would conflict with full participation in the current study or confound the observation or interpretation of the study findings

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in vitamin D status 5 days following supplementation with cholecalciferol | Patients will be followed between the initial preoperative evaluation day and an average duration of 5 days
  Subjects will receive 150,000 IU or 100,000 IU cholecalciferol (vs. placebo) 3-7 days before surgery during their pre-operative assessment. Vitamin D status on the day of pre-operative assessment will be compared to vitamin D status on the day of surgery. To assess vitamin D status, we will measure serum: 1) 25-hydroxyvitamin D; 2) Parathyroid hormone; 3) Vitamin D binding protein; 4) LL-37; 5) Albumin; and 6) Calcium levels.

SECONDARY OUTCOMES:
Change in pre-surgical vitamin D status 1 day after surgery | Patients will be followed between the day of surgery and an average duration of 1 day after surgery
  Subjects will receive either pre-operative supplementation with 150,000 IU or pre-operative supplementation with 100,000 IU cholecalciferol plus 50,000 IU cholecalciferol on post-operative day 1 (vs. placebo). Vitamin D status will be compared between the day of surgery and post-operative day 1. To assess vitamin D status, we will measure: 1) 25-hydroxyvitamin D; 2) Parathyroid hormone; 3) Vitamin D binding protein; 4) LL37; 5) Albumin; and 6) Calcium levels.
Change in pre-surgical vitamin D status 2 weeks after surgery | Patients will be followed between the day of surgery and an average duration of 14 days after surgery
  Subjects will receive either pre-operative supplementation with 150,000 IU or pre-operative supplementation with 100,000 IU cholecalciferol plus 50,000 IU cholecalciferol on post-operative day 1 (vs. placebo). Vitamin D status will be compared between the day of surgery and post-operative day 10-18. To assess vitamin D status, we will measure: 1) 25-hydroxyvitamin D; 2) Parathyroid hormone; 3) Vitamin D binding protein; 4) LL37; 5) Albumin; and 6) Calcium levels.
Change in pre-surgical vitamin D status 3 months after surgery | Patients will be followed between the day of surgery and an average of 90 days after surgery
  Subjects will receive either pre-operative supplementation with 150,000 IU or pre-operative supplementation with 100,000 IU cholecalciferol plus 50,000 IU cholecalciferol on post-operative day 1 (vs. placebo). Vitamin D status will be compared between the day of surgery and post-operative day 80-100. To assess vitamin D status, we will measure: 1) 25-hydroxyvitamin D; 2) Parathyroid hormone; 3) Vitamin D binding protein; 4) LL37; 5) Albumin; and 6) Calcium levels.

OTHER OUTCOMES:
Incidence of post-operative complications within 3 months of surgery | Patients will be followed between the day of surgery and an average of 90 days after surgery
  Subjects will receive either pre-operative supplementation with 150,000 IU or pre-operative supplementation with 100,000 IU cholecalciferol plus 50,000 IU cholecalciferol on post-operative day 1 (vs. placebo). The incidence of post-operative complications will be assessed between the day of surgery and post-operative day 80-100. To assess the incidence of post-surgical complications, we will measure rates of: 1) pneumonia; 2) urinary tract infection; 3) surgical site infection; 5) sepsis/bacteremia; 6) infected hardware; 7) hospital readmission; and 8) mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Sadeq A Quraishi, MD, MMSc, Principal Investigator — Harvard Medical School, Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States